CLINICAL TRIAL: NCT05453786
Title: A Phase 1 Clinical Trial to Compare and Evaluate Safety and Pharmacokinetic Characteristics After Administration of SID1903 (Fixed-dose Combination) or Loose Combination in Healthy Adult Volunteers
Brief Title: A Pharmacokinetic Study of SID1903 (FDC of Dapagliflozin and Sitagliptin) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SID1903_002
Record Dates: First submitted 2022-06-30; First posted 2022-07-12 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-06

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): Period 1: SID1903-R1, SID1903-R2 / Period 2: SID1903
  Interventions: Drug: SID1903; Drug: SID1903-R1/SID1903-R2
- Sequence B (Experimental): - Period 1: SID1903 / Period 2: SID1903-R1, SID1903-R2
  Interventions: Drug: SID1903; Drug: SID1903-R1/SID1903-R2

INTERVENTIONS:
Drug: SID1903 — Single oral administration of SID1903 after an overnight fast
Drug: SID1903-R1/SID1903-R2 — Single oral administration of SID1903-R1 and SID1903-R2 after an overnight fast

SUMMARY:
This study is to compare and evaluate the safety and pharmacokinetic characteristics (PK) after administration of SID1903 and SID1903-R1/SID1903-R2 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged between 19 years and 55 years(inclusive)
* Subjects weighing at least 50.0 kg and no more than 100 kg (inclusive) with a BMI between 18.5 kg/m2 and 30.0 kg/m2 (inclusive)
* Subjects with neither congenital nor chronic diseases requiring treatment, and no abnormal symptoms or findings upon medical examination
* Subjects considered eligible for the study participation in accordance to the results of vital signs, physical examinations, 12-lead ECG, clinical laboratory tests (including hematology, blood chemistry, urinalysis, serology, etc.) and urine drug screening conducted at the time of screening, based on the investigational product (IP) characteristics
* Subjects who has a full understanding in participation of the study, voluntarily provide a written consent in participation, and give full agreement in following the subject guidelines throughout the entire study period

Exclusion Criteria:

* Subjects with any clinically significant hepatic, renal, nervous, respiratory, endocrine, circulatory, genitourinary, cardiovascular, digestive, musculoskeletal systemic diseases, psychosis disorders, or other medical history
* Subjects with a past medical history of gastrointestinal disease or gastrointestinal surgeries
* Pregnant subjects with a positive urine HCG test, or lactating female subjects
* Subjects with hypersensitivity reactions or a clinically significant medical history of hypersensitivity reactions to drug substances and additives containing drug substances or other drugs
* Subjects with clinically significant 12-lead ECG findings
* Subjects with clinically significant laboratory test results as follows: Liver function test (AST, ALT, ALP, γ-GTP and total bilirubin), Creatinine, eGFR
* Subjects with a past history of drug abuse or a positive urine drug test
* Subjects with SBP ≥ 140 mmHg or ≤ 90 mmHg; DBP ≥ 90 mmHg or ≤ 60 mmHg; PR ≤ 50 beats/min or ≥ 100 beat/min
* Subjects following an unusual diet or consumption of food which may affect the absorption, distribution, metabolism and excretion of the IP
* Subjects taking drugs known to significantly induce or inhibit drug metabolizing enzymes, including barbitals prior to the first IP administration
* Subjects who have participated and were given any other study drugs in other clinical study within 6 months prior to the first IP administration
* Subjects who have consistently drunk alcohol within 6 months
* Subjects who have smoked more than 10 cigarettes/day on average
* Subjects who have done and are unable to refrain from strenuous activity
* Subjects who are planning for pregnancy or not willing to use a medically reliable forms of contraception
* Subjects otherwise considered ineligible for participation due to other reasons including clinical laboratory test results not mentioned in the inclusion/exclusion criteria at the investigator's discretion

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
AUC0-t | up to 72hours
Cmax | up to 72hours

SECONDARY OUTCOMES:
Tmax | up to 72hours
AUCinf | up to 72hours
t1/2 | up to 72hours
CL/F | up to 72hours
Vd/F | up to 72hours
λz | up to 72hours
MRT | up to 72hours

CONTACTS AND LOCATIONS:
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lukka PB, Tang W, Hammarstedt A, Conrad T, Heijer M, Karlsson C, Boulton DW. Racial Comparison of the Pharmacokinetics and Safety of Fixed-dose Combination of Dapagliflozin/Sitagliptin in Western and Korean Healthy Adults. Clin Ther. 2024 Sep;46(9):717-725. doi: 10.1016/j.clinthera.2024.07.007. Epub 2024 Aug 23. PMID 39179458